CLINICAL TRIAL: NCT02873832
Title: Efficacy of Heat-shock Protein (HSP) Inhibitors in Myeloproliferative Syndromes (MPS): Fundamental Observational in Vitro Study Using Samples From a Collection
Brief Title: Efficacy of Heat-shock Protein (HSP) Inhibitors in Myeloproliferative Syndromes (MPS)
Acronym: HSP-SMP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GIRODON 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Myeloproliferative Syndrome
MeSH Terms: interventions — Blood Specimen Collection; Flow Cytometry; Blotting, Western

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- MPS
  Interventions: Biological: Blood sample; Other: Flow cytometry; Other: western blot
- Control
  Interventions: Biological: Blood sample; Other: Flow cytometry; Other: western blot

INTERVENTIONS:
Biological: Blood sample
Other: Flow cytometry
Other: western blot

SUMMARY:
Heat-shock proteins (HSP) have been very highly conserved throughout the evolution of species and are characterized by their chaperone function, thanks to their ability to prevent aggregation and to promote the renaturation/break down of damaged proteins. Among other targets, they also chaperone JAK2, a key step that is deregulated in signalling in myeloproliferative syndromes (MPS) because of the JAK2V617F mutation. These HSP also have a potent cytoprotective action through their multiples inhibiting effects on apoptotic processes.

Little is known about levels of HSP expression, in particular for HSP70 and HSP27, in MPS cells.

However, in vitro studies of different cell models have shown the interest of HSP90 inhibitors in slowing cell proliferation in MPS. These results have been confirmed in animal models with results in terms of blood counts and overall survival. In addition, it seems that the V617F mutated form of JAK2 is more sensitive than the wild-type to HSP90 inhibitors. Finally, inhibitors of HSP90 remain efficacious with regard to the inhibition of cell growth, even in cases of resistance to JAK2 inhibitors. Nonetheless, HSP90 inhibitors are known to stimulate the expression of other HSP, notably HSP27 and HSP70, which are, through their properties, tumorigenic and could lead to an escape phenomenon. Thus the combined use of several HSP inhibitors could be beneficial, and eventually present synergistic effects on the inhibition of tumour processes.

ELIGIBILITY:
Inclusion Criteria:

MPS Patients:

* Patients with MPS
* Patients who have been informed and not objected to the tests
* Patients over 18 years old
* Patients whose samples have been preserved at the CRB in the "Haemopathies" collection

Control patients:

* Patients over 18 years old
* Pregnant patients
* Patients who have been informed and not objected to the collection of their cord blood after the delivery

Exclusion Criteria:

* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myeloproliferative Syndrom
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparing the level of expression of HSP (HSP90, HSP70, HSP27) between cells from a collection of samples of patients with myeloproliferative disease and healthy controls . | through study completion, an average of 1 year
  Level of protein expression using flow cytometry and western blot

SECONDARY OUTCOMES:
Cell death after in vitro treatment with different HSP inhibitors | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France